CLINICAL TRIAL: NCT04703387
Title: Prospective Observational Study on Left Ventricular Diastolic Dysfunction as a Predictor of Weaning Failure From Mechanical Ventilation
Brief Title: Left Ventricular Diastolic Dysfunction as a Predictor of Weaning Failure From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Azzam Abdellatif Elsayed, Dr, Tanta University
Other Study IDs: 33855/6/20
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Left Ventricular Diastolic Dysfunction; Weaning Failure; Mechanical Ventilation Complication; Diaphragmatic Disorder
Keywords: Mechanical Ventilation Complication; Left Ventricular Diastolic Dysfunction; Pulmonary Edema; echocardiography
MeSH Terms: conditions — Ventricular Dysfunction, Left; Pulmonary Edema | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postextubation Success
  Interventions: Diagnostic Test: transthoracic echocardiography
- Postextubation Distress
  Interventions: Diagnostic Test: transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — Trans-mitral flow velocities (peak early diastolic E and peak late diastolic A) will be recorded with pulsed-wave Doppler, placing the sample volume at the mitral valve tips from the apical 4-chamber view; deceleration time of the E wave (DTE) will be measured. Peak early diastolic velocity will be obtained with tissue Doppler imaging (TDI), in the apical 4-chamber view, positioning the pulsed-wave Doppler sample volume at or 1 cm within the septal insertion sites of the mitral leaflets, so as to cover the longitudinal excursion of the mitral annulus in both systole and diastole. Then, the E/A ratio and the trans-mitral inflow E wave to mitral annular e' (E/e) will be calculated.Diaphragmatic thickness will be assessed in the zone of apposition of the diaphragm to the rib cage between the 8th and 10th intercostal spaces using a 3-12 MHz linear array probe , we will record changes in diaphragm vertical excursion using M-mode ultrasound.
  Other Names: diaphragm ultrasonographic

SUMMARY:
Both premature and delayed extubation prolong the duration of mechanical ventilation and the intensive care unit (ICU) length of stay and increase morbidity and mortality. Therefore, accurate prediction of postextubation distress and the early diagnosis of the causes responsible for failure of a trial of pressure support ventilation are of paramount importance to improve the outcome of mechanically ventilated patients in the ICU.

This observational study is designed to test the ability of cardiac and diaphragm function assessed by bedside ultrasound to predict extubation failure within 48 h and re-intubation within 1 week after extubation.

DETAILED DESCRIPTION:
Weaning from mechanical ventilation is the process of gradual ventilatory support reduction to the patient subjected to mechanical ventilation for more than 24 hours. Determining the correct time to extubate mechanically ventilated patients is a crucial issue in the critical care practice.

Spontaneous breathing trial (SBT) is recommended to predict weaning outcome. However, 13% to 26% of patients who are extubated following a successful SBT need to be reintubated within 48 hours.

Traditional indicators, such as respiratory rate (RR), minute ventilation, tidal volume (VT), and the rapid shallow breathing index (RSBI), can reflect patients' integral conditions, but none has shown great prognostic accuracy for weaning failure.

Although there are several causes of weaning failure, cardiac function deterioration during the weaning process combined with acute pulmonary edema is considered the leading cause of weaning failure. The transition from positive to negative thoracic pressure increases venous return and left ventricular afterload, decreases left ventricular compliance and may induce cardiac ischemia. All of these factors tend to increase ventricular filling pressures and may consequently lead to weaning-induced pulmonary edema. The efficacy of echocardiography for predicting weaning failure has been reported, however there is debate over the predictive value of echocardiography in this setting continues due to differences in weaning technique and outcome evaluation.

The diaphragm is the principal respiratory muscle. With an excursion of 1 to 2 cm, it provides nearly 75% of the resting pulmonary ventilation, while during the forced breathing, its amplitude is up to 7 to 11 cm. However, the diaphragm is vulnerable to damage from hypotension, hypoxia, and sepsis, which are very common in critically ill patients. While in surgical patients, diaphragm dysfunction is often caused by acute insults such as trauma or surgical procedures. In addition, mechanical ventilation itself can decrease the force of the diaphragm and induce diaphragmatic dysfunction, named as ventilator-induced diaphragmatic dysfunction. Many studies have shown that Diaphragm dysfunction is responsible for a number of pulmonary complications, including atelectasis and pneumonia, which are risk factors for extubation failure. and might lead to weaning failure and long-term mechanical ventilation.

Some studies have reported that diaphragmatic excursion (DE) or and diaphragmatic thickening fraction (DTF) could predict extubation failure.

Although transthoracic echocardiography and diaphragm ultrasound have been confirmed in independently assessing extubation outcomes, few studies have shown their different roles in the weaning process until now.

ELIGIBILITY:
• Inclusion criteria: All patients aged more than 40 years who are intubated and mechanically ventilated for more than 48 hours, with improvement of underlying cause of acute respiratory failure and considered ready to undergo a spontaneous breathing trial (SBT) by the attending physician on the basis of readiness-to-wean criteria used in our surgical ICUn Criteria

-

Exclusion Criteria:

1. Planning for tracheostomy after the SBT.
2. Severe mitral stenosis, severe regurgitation, or prosthetic mitral valve.
3. History of diaphragmatic dysfunction as diaphragmatic palsy, cervical spine injury, or neuromuscular disease.
4. Pneumothorax or pneumo-mediastinum.
5. Use of muscle-paralyzing agents within 48 h before the study.
6. Poor echocardiographic windows or difficult windows of diaphragmatic movement as women in late pregnancy or obese patients.
7. Extubation failure definitely caused by upper airway obstruction.
8. Planned prophylactic noninvasive ventilation (NIV) after extubation.
9. Atrial fibrillation or atrioventricular conduction abnormality.

   -

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged more than 40 years who are intubated and mechanically ventilated for more than 48 hours, with improvement of underlying cause of acute respiratory failure and considered ready to undergo a spontaneous breathing trial (SBT) by the attending physician on the basis of readiness-to-wean criteria used in our surgical ICUn Criteria
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Weaning failure | within 48 hours after extubation
  Weaning failure predicted by diastolic dysfunction assessed by E/Ea.

SECONDARY OUTCOMES:
Weaning failure | within 48 hours after extubation
  Weaning failure predicted by Diaphragmatic function assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided